CLINICAL TRIAL: NCT00712309
Title: Endovascular Treatment of Atherosclerotic Popliteal Artery Lesions - Balloon Angioplasty Versus Primary Stenting
Brief Title: Endovascular Treatment of Popliteal Artery - Balloon Angioplasty Versus Primary Stenting
Acronym: ETAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Herz-Zentrums Bad Krozingen (Other)
Collaborators: University Hospital Tuebingen (Other); Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Thomas Zeller, MD, Herzzentrums Bad Krozingen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ETAP Protocol 2.0
Record Dates: First submitted 2008-07-08; First posted 2008-07-09 (Estimated); Last update posted 2009-02-10 (Estimated); Status verified 2009-02

CONDITIONS: Popliteal Artery
Keywords: atherosclerotic; lesions
MeSH Terms: interventions — Angioplasty, Balloon

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Percutaneous transluminal angioplasty (PTA)
  Interventions: Device: balloon-angioplasty (PTA)
- 2 (Active Comparator): Primary stenting
  Interventions: Device: Lifestent

INTERVENTIONS:
Device: Lifestent — Stent for endovascular treatment of popliteal artery lesions
  Arms: 2
Device: balloon-angioplasty (PTA) — PTA for endovascular treatment of popliteal artery lesions
  Arms: 1

SUMMARY:
1. Does primary stenting have a lower 12-month restenosis rate than PTA alone in the treatment of atherosclerotic lesions of the popliteal artery?

   * Alternative hypothesis: "Primary stenting with the Edwards LifeStent is associated with a lower restenosis rate than PTA alone in patients with atherosclerotic lesions of the popliteal artery at 12 months"
   * Null hypothesis: "Primary stenting with the Edwards LifeStent is not associated with a lower 12-month restenosis rate than PTA alone in patients with atherosclerotic lesions of the popliteal artery""
2. Does comparison of the two intervention groups (PTA alone, stenting) disclose differences in terms of the secondary endpoints?
3. How do the intervention methods compare in terms of safety/incidence of adverse effects?
4. What are the long-term clinical implications of the two treatment methods?

ELIGIBILITY:
Inclusion Criteria:

* The patient is at least 21 years old
* The patient or legal representative provided written informed consent
* The patient agrees to comply with the protocol-mandated follow-up visits and testing regime
* The patient has lifestyle-limiting claudication or critical limb ischemia defined as: Fontaine stage IIa-IV/ Rutherford 1-5 category
* The target lesion located within the popliteal artery has angiographic evidence of stenosis > 70% or occlusion (by visual estimate)
* At least one vessel runoff to the foot
* The patient has no other relevant inflow or outflow stenosis (> 50%), however when needed iliac or femoral intervention may be done during study procedure.

Exclusion Criteria:

* The patient is currently participating in a drug or another device study.
* The popliteal artery target lesion has previously been subintimal recanalized
* The patient has a history of bleeding diatheses or coagulopathy
* Female patients that are pregnant
* The patient has a contraindication (including allergic reaction) to platelet aggregation inhibitors or heparin
* The patient is unable to conform to the study protocol follow-up procedures or visits.
* The patient has a life expectancy of <24 months
* The patient has concomitant renal failure which requires dialysis
* The patient has a contraindication (including allergic reaction) to or a known sensitivity to contrast media
* The duplex ultrasound/angiography of the target lesion must NOT meet the following criteria:

  * The popliteal artery target lesion stenosis/occlusion is also continuously located within the superficial femoral artery and/or tibiofibular tract
  * The popliteal artery target lesion is restenotic
  * The popliteal artery has been subintimal recanalized

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2007-02; Primary Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Restenosis rate (duplex ultrasound or angiographic stenosis >50% of vascular lumen diameter; PVR > 2.4 m/s) | 12-month

SECONDARY OUTCOMES:
Primary patency | 12 and 24 months

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Herzzentrum Bad Krozingen, Bad Krozingen
  - Universitäres Herzzentrum Hamburg, Hamburg

REFERENCES:
- [Derived] Rastan A, Krankenberg H, Baumgartner I, Blessing E, Muller-Hulsbeck S, Pilger E, Scheinert D, Lammer J, Beschorner U, Noory E, Neumann FJ, Zeller T. Stent placement vs. balloon angioplasty for popliteal artery treatment: two-year results of a prospective, multicenter, randomized trial. J Endovasc Ther. 2015 Feb;22(1):22-7. doi: 10.1177/1526602814564386. PMID 25775675
- [Derived] Rastan A, Krankenberg H, Baumgartner I, Blessing E, Muller-Hulsbeck S, Pilger E, Scheinert D, Lammer J, Gissler M, Noory E, Neumann FJ, Zeller T. Stent placement versus balloon angioplasty for the treatment of obstructive lesions of the popliteal artery: a prospective, multicenter, randomized trial. Circulation. 2013 Jun 25;127(25):2535-41. doi: 10.1161/CIRCULATIONAHA.113.001849. Epub 2013 May 21. PMID 23694965